CLINICAL TRIAL: NCT00225017
Title: Switch to Atazanavir and Brachial Artery Reactivity (SABAR) Study: Endothelial Function in HIV-Infected Subjects Switched to an Atazanavir Regimen
Brief Title: Switch to Atazanavir and Brachial Artery Reactivity (SABAR) Study
Acronym: SABAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Robert L. Murphy, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SABAR
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infection; Hyperlipidemia
Keywords: Atazanavir; Endothelial function; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hyperlipidemias | interventions — Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): ARM A: Switch current PI to atazanavir 400 mg once daily plus current > 2 nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) for 24 weeks.
  Subjects currently on ritonavir (RTV) (400 mg BID or greater) or RTV-boosted PI (<400 mg/day) , or tenofovir (TDF) as backbone NRTI therapy, will switch to ATV 300 mg boosted with RTV 100mg once daily.
  Interventions: Drug: Atazanavir
- B (Active Comparator): ARM B: Continue current antiretroviral regimen (single or RTV-boosted PI plus > 2 NRTIs) for 24 weeks
  Interventions: Drug: current antiretroviral regimen

INTERVENTIONS:
Drug: Atazanavir — atazanavir 400 mg once daily
  Other Names: Reyataz
  Arms: A
Drug: current antiretroviral regimen — Continue current antiretroviral regimen for 24 weeks, single or RTV-boosted PI plus > 2 NRTIs
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the change in brachial artery reactivity in HIV-infected subjects with elevated lipid levels who are switched to an atazanavir containing antiretroviral regimen

DETAILED DESCRIPTION:
HIV-infected subjects on a stable protease inhibitor (PI) containing antiretroviral regimen with plasma HIV RNA <500 copies/mL, who have LDL cholesterol levels >130 mg/dL or fasting triglycerides levels >200 mg/dL, will be randomized (1:1) to continue their current antiretroviral regimen or to switch the PI to atazanavir (ATV). Brachial artery reactivity will be measured before (at entry) and 12 and 24 weeks after subjects are randomized.

ARM A: Switch current PI to atazanavir 400 mg once daily plus current > 2 nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) for 24 weeks.

Subjects currently on ritonavir (RTV) (400 mg BID or greater) or RTV-boosted PI (<400 mg/day) , or tenofovir (TDF) as backbone NRTI therapy, will switch to ATV 300 mg boosted with RTV 100mg once daily.

ARM B: Continue current antiretroviral regimen (single or RTV-boosted PI plus > 2 NRTIs) for 24 weeks

Brachial artery reactivity in response to two vasoactive stimuli (increased forearm blood flow and nitroglycerin) will be assessed by measuring brachial artery diameter.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* HIV-1 RNA < 500 copies/ml
* Fasting LDL cholesterol >130 mg/dl OR fasting triglycerides >200 mg/dl
* CD4 count >100 cells/mm
* Stable antiretroviral regimen for at least 12 weeks prior to study entry that includes a protease inhibitor (PI) with or without ritonavir boosting

Exclusion Criteria:

* History of heart disease, uncontrolled hypertension, peripheral vascular disease
* Current non-nucleoside reverse transcriptase inhibitor (NNRTI) in the PI-containing regimen within 4 weeks
* Prior or current use of atazanavir
* Initiation of treatment with lipid-lowering drugs within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Murphy, MD, Study Chair — Northwestern University; James H Stein, MD, Study Chair — University of Wisconsin, Madison
Locations (7):
- United States (5):
  - University of California, San Diego, California
  - Northwestern Universtiy, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Cincinnati, Cincinnati, Ohio
  - University of Wisconsin, Madison, Wisconsin
- ACLIRES - Argentina S.R.L., Buenos Aires, Argentina
- Universita degli studi di Modena e Reggio Emilia, Modena, Italy

REFERENCES:
- [Result] Murphy RL, Berzins B, Zala C, Fichtenbaum C, Dube MP, Guaraldi G, Torriani F, Belsey E, Mitchell C, Stein JH; SABAR Study Team. Change to atazanavir/ritonavir treatment improves lipids but not endothelial function in patients on stable antiretroviral therapy. AIDS. 2010 Mar 27;24(6):885-90. doi: 10.1097/QAD.0b013e3283352ed5. PMID 19952712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period June 2005 to November 2007 at four clinics in the United States, one in Italy, and one in Argentina
Groups:
- Atazanavir Switch: ARM A: Switch current PI to atazanavir 400 mg once daily plus current > 2 nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) for 24 weeks.
  Subjects currently on ritonavir (RTV) (400 mg BID or greater) or RTV-boosted PI (<400 mg/day) , or tenofovir (TDF) as backbone NRTI therapy, will switch to ATV 300 mg boosted with RTV 100mg once daily.
- Control (Continue Protease Inhibitor): ARM B: Continue current antiretroviral regimen (single or RTV-boosted PI plus > 2 NRTIs) for 24 weeks
Period: Overall Study
Arm/Group | Atazanavir Switch | Control (Continue Protease Inhibitor)
Started | 26 | 24
Completed | 26 | 23 (1 subject did not complete week 24 assessments)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atazanavir Switch | Control (Continue Protease Inhibitor) | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 50
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Full Range); unit: years] | 43 [25 to 68] | 43 [33 to 58] | 43 [25 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 22 | 20 | 42
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32
  Argentina | 8 | 7 | 15
  Italy | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Brachial Artery Flow Mediated (FMD) Vasodilation Between Arms From Baseline to Week 24
Description: Brachial artery reactivity assessed by noninvasively measuring brachial artery diameter and flow velocities in response to overinflated blood pressure cuff (Flow mediated dilation (FMD))in subjects switching to atazanavir and in subjects continuing on a stable antiretroviral regimen
Time Frame: Baseline to week 24
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Atazanavir Switch | Control (Continue Protease Inhibitor)
Number analyzed (Participants) | 26 | 23
percentage change | -1.14 [-2.24 to 1.63] | 0.25 [-1.58 to 1.84]
Statistical Analysis 1: Comparison: Atazanavir Switch vs Control (Continue Protease Inhibitor); Test type: Non-Inferiority or Equivalence — 25 subjects per arm will have 80% power to detect a difference between groups in mean FMD change of 2.9%, and 90% power to detect a mean FMD change of 3.4%; p = 0.601, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.384, 95% CI 2-sided [-2.080 to 1.312], Standard Deviation 1

2. Secondary Outcome: Change in Total Cholesterol Levels From Baseline to Week 24
Description: Total cholesterol level changes within and between arms
Time Frame: Baseline to 24 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Atazanavir Switch | Control (Continue Protease Inhibitor)
Number analyzed (Participants) | 26 | 23
mg/dL | -25 [-46 to -14] | 2 [-25 to 31]
Statistical Analysis 1: Comparison: Atazanavir Switch vs Control (Continue Protease Inhibitor); Test type: Superiority or Other; p < 0.009, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Changes in LDL Particle Number From Baseline to Week 24
Description: Change in LDL particle number
Time Frame: Baseline to 24 weeks
Measure: Median (Inter-Quartile Range); unit: nmol/l
Arm/Group | Atazanavir Switch | Control (Continue Protease Inhibitor)
Number analyzed (Participants) | 26 | 23
nmol/l | -194 [-387 to 26] | -116 [-335 to 84]
Statistical Analysis 1: Comparison: Atazanavir Switch vs Control (Continue Protease Inhibitor); Test type: Superiority or Other; p = 0.141, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Atazanavir Switch | Control (Continue Protease Inhibitor)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No